CLINICAL TRIAL: NCT04471844
Title: EF-32: Pivotal, Randomized, Open-Label Study of Optune® (Tumor Treating Fields, 200kHz) Concomitant With Radiation Therapy and Temozolomide for the Treatment of Newly Diagnosed Glioblastoma
Brief Title: Pivotal, Randomized, Open-label Study of Optune® (Tumor Treating Fields) Concomitant With RT & TMZ for the Treatment of Newly Diagnosed GBM
Acronym: EF-32
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIDENT EF-32
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Randomly assigned equally to one of two groups:
  1. Treatment arm I: Patients receive TTFields at 200 kHz to the brain using the Optune® System together with RT and TMZ, followed by maintenance TMZ concomitant with the Optune® treatment.
  2. Treatment arm II: Patients receive RT and TMZ alone, followed by maintenance TMZ concomitant with TTFields at 200 kHz to the brain using the Optune®.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Optune® + RT + TMZ for 6 weeks (Experimental): Optune® + RT + TMZ for 6 weeks, followed by Optune® + TMZ until the tumor progresses. Optune treatment is maintained until second disease progression.
  Interventions: Device: Optune®
- RT +TMZ for 6 weeks (Active Comparator): RT +TMZ for 6 weeks followed by Optune® + TMZ until the tumor progresses. Optune treatment is maintained until second disease progression.
  Interventions: Device: Optune®

INTERVENTIONS:
Device: Optune® — Optune® is a commercial, portable, battery-operated device intended for continuous home use, which delivers TTFields at a frequency of 200kHz to the brain by means of insulated transducer arrays. The Optune® device produces electric forces intended to disrupt cancer cell division.
  In treatment arm I, the patient starts Optune® concurrently with RT/TMZ for 6 weeks, followed by Optune® + TMZ until second disease progression.
  In treatment arm II, the patient starts RT/TMZ for 6 weeks, followed by Optune® + TMZ until second disease progression.

SUMMARY:
To test the effectiveness and safety of Optune® given concomitantly with radiation therapy (RT) and temozolomide (TMZ) in newly diagnosed GBM patients, compared to radiation therapy and temozolomide alone. In both arms, Optune® and maintenance temozolomide are continued following radiation therapy.

DETAILED DESCRIPTION:
Optune® is a medical device that has been approved for the treatment of recurrent and newly diagnosed glioblastoma (GBM) by the Food and Drug Administration (FDA) in the United States. Optune® has obtained a CE mark in Europe for recurrent and newly diagnosed GBM.

The current standard of care for GBM includes the addition of Optune® to maintenance temozolomide (TMZ), following the completion of radiation therapy (RT).

The purpose of the current study is to test if the earlier introduction of Optune®, at the time of radiation therapy (which is given together with temozolomide), improves clinical outcomes compared to the standard of care.

The study will randomize 950 subjects equally to one of two treatment arms:

1. Treatment arm I: Patients receive TTFields at 200 kHz to the brain using the Optune® System together with RT and TMZ, followed by maintenance TMZ concomitant with the Optune® treatment.
2. Treatment arm II: Patients receive RT and TMZ alone, followed by maintenance TMZ concomitant with TTFields at 200 kHz to the brain using the Optune®.

All patients are to receive standard RT and TMZ treatment followed by maintenance TMZ chemotherapy and Optune® according to the current standard of care regimen.

Optune® will continue until second disease progression per 2010 RANO Criteria unless any of the treatment discontinuation conditions described under criteria for patient withdrawal or termination are met.

After surgery or biopsy, subjects that would like to participate will be required to submit samples of their tumor to a lab for testing. The results of this test will be used for randomization into the trial.

If the subject is assigned to the treatment group that will start Optune® therapy during radiation therapy, Optune® therapy will begin within 10 days of enrolling in the study and no later than the first day of RT and TMZ treatment.

After the initial visit, subjects will continue treatment at home, while pursuing normal daily routines. Subjects are required to use the device for at least 18 hours a day. Short breaks in treatment for personal hygiene and other personal needs is allowed. Total usage time will be recorded and provided to the site and sponsor.

Subjects will be required to return to the clinic per the study protocol.

After the second disease progression, subjects will return to the clinic for one final visit approximately 30 days after the last treatment with Optune® or after second disease progression, the latter of the two per protocol.

After completing active participation in the study, subjects will be contacted once per month to answer basic questions about their health status.

ELIGIBILITY:
*Age Limits - 18 years or older outside of the US, 22 years or older within the US.

Inclusion Criteria:

1. Histologically confirmed diagnosis of GBM according to WHO 2016 classification criteria.
2. Age ≥ 22 years in US and Age ≥ 18 years in Ex-US
3. Recovered from maximal debulking surgery, if applicable (gross total resection, partial resection, and biopsy-only patients are all acceptable)
4. Planned treatment with RT/TMZ followed by TTFields and maintenance TMZ (150-200 mg/m2 daily x 5 d, q28 days)
5. Karnofsky performance status ≥ 70
6. Life expectancy ≥ least 3 months
7. Participants of childbearing age must use highly effective contraception. An effective method of birth control is defined as one that results in a failure rate of less than 1% per year when used consistently and correctly. The Investigator must approve the selected method, and may consult with a gynecologist as needed.
8. All patients must understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.
9. Stable or decreasing dose of corticosteroids for the last 7 days prior to randomization, if applicable.
10. Concomitant RT with TMZ treatment planned to start no later than 8 weeks from surgery
11. Women of childbearing potential must have a negative β-HCG pregnancy test documented within 14 days prior to randomization
12. Is able to have MRI with contrast of the brain

Exclusion Criteria:

1. Progressive disease (per investigator's assessment)
2. Infratentorial or leptomeningeal disease
3. Participation in another clinical treatment study during the pre-treatment and/or the treatment phase of the study
4. Pregnancy or breast-feeding.
5. Significant co-morbidities at baseline which would preclude maintenance RT or TMZ treatment, as determined by the investigator:

   1. Thrombocytopenia (platelet count < 100 x 103/μL)
   2. Neutropenia (absolute neutrophil count < 1.5 x 103/μL)
   3. CTC grade 4 non-hematological Toxicity (except for alopecia, nausea, vomiting)
   4. Significant liver function impairment - AST or ALT > 3 times the upper limit of normal
   5. Total bilirubin > 1.5 x upper limit of normal
   6. Significant renal impairment (serum creatinine > 1.7 mg/dL, or > 150 µmol/l)
   7. History of any psychiatric condition that might impair patient's ability to understand or comply with the requirements of the study or to provide consent
6. Implanted pacemaker, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
7. Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness)
8. History of hypersensitivity reaction to TMZ or a history of hypersensitivity to DTIC.
9. Additional malignancies that are progressing or required active treatment in the last two years.
10. Admitted to an institution by administrative or court order.
11. Known allergies to medical adhesives or hydrogel
12. A skull defect (such as, missing bone with no replacement)
13. Prior radiation treatment to the brain for the treatment of GBM
14. Any serious surgical/post-operative condition that may put the participant at risk according to the investigator.
15. Standard TTFields exclusion criteria include

    1. Active implanted medical devices
    2. Bullet fragments
    3. Skull defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 981 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5 years
  Survival will be measured from the time of randomization until date patient is alive.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 5 years
  PFS will be measured from the date of randomization to the date of progression based on the 2010 RANO Criteria.
1- and 2-year survival rates | 5 years
  The analyses will be performed based on estimated proportions of patients who are on study at 12 and 24 months in both arms of the study.
Overall Radiological response (ORR) | 5 years
  The analyses will be performed based on the 2010 RANO criteria, and comparison between the rates of response.
Next progression-free survival (PFS2) | 5 years
  PFS2 will be measured from the time of randomization to second tumor progression.
Progression-free survival at 6 (PFS6) and 12 months (PFS12) | 5 years
  The analyses will be estimated proportions of patients who are progression-free at 6 and 12 months in both arms of the study.
Severity and frequency of adverse events | 5 years
  The analyses will be performed based on the incidence, severity, frequency of adverse events, and their association with study treatments.
Quality of Life EORTC Questionnaire | 5 years
  The analyses will be assessed using the EORTC QLQ C-30 questionnaire with BN-20 (brain symptom) supplement.
The NANO scale | 5 years
  The Neurological assessment in Neuro-Oncology will be assessed using the NANO scale questionnaire and per the 2010 RANO criteria.

CONTACTS AND LOCATIONS:
Locations (133):
- United States (87):
  - Grandview Cancer Center, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic- Arizona, Phoenix, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Providence St. Joseph Medical Center and The Roy and Patricia Disney Family Cancer Center, Burbank, California
  - City of Hope National Medical Center, Duarte, California
  - TRIO - St. Jude Heritage Healthcare/St. Jude Medical Center, Fullerton, California
  - University of California at San Diego - Moores Cancer Center, La Jolla, California
  - Norris Comprehensive Cancer Center at USC, Los Angeles, California
  - Cedars - Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital - Hoag Cancer Center, Newport Beach, California
  - St. Joseph Hospital of Orange, Orange, California
  - University of California - Irvine/UCI Medical Center, Orange, California
  - Stanford University Cancer Institute, Palo Alto, California
  - Sharp Memorial Hospital - X-Ray Medical Group Radiation Oncology, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - John Wayne Cancer Institute at St. John's Health Center, Santa Monica, California
  - University of Colorado Cancer Center Anschutz, Aurora, Colorado
  - HCA Research Institute - Blue Sky Neurology - Denver, Englewood, Colorado
  - Hartford Healthcare Medical Group - Hartford Hospital The Gray Cancer Center, Hartford, Connecticut
  - Lynn Cancer Institute, Marcus Neuroscience Institute, Boca Raton, Florida
  - Baptist Health - Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - AdventHealth, Orlando, Florida
  - Orlando Health UF Health Cancer Center, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Inc, Tampa, Florida
  - Piedmont Healthcare Brain Tumor Center, Atlanta, Georgia
  - The Emory Clinic - Emory Healthcare - Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Inc., Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Parkview Cancer Institute - Fort Wayne Radiation Oncology Associates, Fort Wayne, Indiana
  - The University of Kansas Cancer Center, Topeka, Kansas
  - University of Louisville - James Graham Brown Cancer Center, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Mary Bird Cancer Center Neuromedical Center, Baton Rouge, Louisiana
  - LSU Health Sciences Center, New Orleans, New Orleans, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - Maine Medical Partners Neurology - Neurosurgery & Spine Associates, South Portland, Maine
  - John Hopkins School of Medicine, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Abbott Northwestern Hospital - Givens Brain Tumor Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel Cancer Center, Columbia, Missouri
  - Health Midwest Ventures Group, Inc - Sarah Cannon HCA Midwest Brain and Spine, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - JFK Neuroscience Institute, HMH JFK University Medical Center, Edison, New Jersey
  - Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Northwell Health System Brain Tumor Center, Lake Success, New York
  - NYU Langone - Laura & Issac Perimutter Cancer Center, New York, New York
  - Mount Sinai - Icahn School of Medicine, New York, New York
  - New York Presbyterian - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina Brain Tumor Program - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Cancer Institute Radiation Oncology, Charlotte, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Forsyth Medical Center-Novant Health, Winston-Salem, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - The James Cancer Hospital and Solove Research Institute - Arthur G James Cancer Hospital, Columbus, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Neuroscience Center, Philadelphia - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny Health Network Cancer Institute, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - MUSC Radiation Oncology Brain & Spine Tumor Program, Charleston, South Carolina
  - SCRI - Tennessee Oncology, Chattanooga, Tennessee
  - West Cancer Center - Germantown, Germantown, Tennessee
  - SCRI - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology Midtown - Austin Brain Tumor Center, Austin, Texas
  - Baylor Charles A. Sammons Cancer Center - Baylor University Medical Center, Dallas, Texas
  - John Peter Smith Health Network - JPS Cancer Center, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - UT Health Mischer Neuroscience - Memorial Herman - UT Neurosciences, Houston, Texas
  - Baylor Scott & White Medical Center, Temple, Texas
  - The University of Vermont Medical Center - University of Vermont Cancer Center, Burlington, Vermont
  - Massey Cancer Center - VCU Medical Center, Richmond, Virginia
  - UW Medical Center - Alvord Brain Tumor Center, Seattle, Washington
  - Swedish Health Services, Seattle, Washington
  - West Virginia University Cancer Institute, Morgantown, West Virginia
- Austria (3):
  - Innsbruck University Hospital, Innsbruck
  - Kepler University Hospital, Linz
  - University Hospital Salzburg, Salzburg
- Belgium (2):
  - Hospital Erasme, Brussels
  - University Hospital Liege - Sart Tilman, Liège
- Canada (7):
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - Nova Scotia Health Authority, Sydney, Nova Scotia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sunnybrook Research Institute - Odette Cancer Centre, Toronto, Ontario
  - CHUM Centre de Recherche, Montreal, Quebec
  - Universite de Sherbrooke - Sherbrooke Centre Hospitalier Universita, Sherbrooke, Quebec
- Czechia (3):
  - Masaryk Memorial Cancer Institute, Brno
  - University Hospital Plzeň, Pilsen
  - Na Homolce Hospital, Prague
- France (8):
  - Institut de cancérologie de l'Ouest, Angers
  - Pierre Wertheimer Hospital, Bron
  - Hôpital la Timone, Marseille
  - University Hospital Nice, Nice
  - Pitié-Salpêtrière University Hospital, Paris
  - Institut de cancérologie de l'Ouest, Saint-Herblain
  - University Institute Cancer Toulouse Oncopole, Toulouse
  - Gustave Roussy Institute, Villejuif
- Germany (6):
  - Charité Campus Virchow Clinic, Berlin
  - University Hospital Essen, Essen
  - University Medical Center Freiburg, Freiburg im Breisgau
  - University Hospital Leipzig, Leipzig
  - Rechts der Isar Hospital, Munich
  - University Hospital Tübingen, Tübingen
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center - Ein Kerem, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (5):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Kyorin University Hospital, Mitaka-shi, Tokyo-To
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo-To
- Switzerland (2):
  - Lausanne University Hospital, Lausanne
  - University Hospital Zurich, Zurich
- United Kingdom (5):
  - Clatterbridge Cancer Centre, Liverpool
  - Guy's Hospital, London
  - Charing Cross Hospital, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Royal Preston Hospital, Preston

REFERENCES:
- [Derived] Miller R, Niazi M, Russial O, Poiset S, Shi W. Tumor treating fields with radiation for glioblastoma: a narrative review. Chin Clin Oncol. 2022 Oct;11(5):40. doi: 10.21037/cco-22-90. PMID 36336899
- [Derived] Miller R, Song A, Ali A, Niazi M, Bar-Ad V, Martinez N, Glass J, Alnahhas I, Andrews D, Judy K, Evans J, Farrell C, Werner-Wasik M, Chervoneva I, Ly M, Palmer J, Liu H, Shi W. Scalp-Sparing Radiation With Concurrent Temozolomide and Tumor Treating Fields (SPARE) for Patients With Newly Diagnosed Glioblastoma. Front Oncol. 2022 Apr 29;12:896246. doi: 10.3389/fonc.2022.896246. eCollection 2022. PMID 35574391